CLINICAL TRIAL: NCT03622632
Title: Pilot Study to Measure Uric Acid in Traumatized Patients: Determinants and Prognostic Association
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Emmanuel Charbonney, MD PhD, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Other Study IDs: 263425
Record Dates: First submitted 2018-07-24; First posted 2018-08-09 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Trauma; Inflammation
Keywords: uric acid; organ failure
MeSH Terms: conditions — Wounds and Injuries; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this project, is to better understand the fluctuation of the level of uric acid in traumatized patients by making serial measurements during their hospitalization in the intensive care unit. In addition, the determinants (e.g. type of trauma, diseases, interventions) of the blood level of uric acid and its association with the development of organ failure will be sought.

ELIGIBILITY:
Inclusion Criteria:

* Direct admission to trauma center
* ≤ 3h after trauma
* ISS ≥ 16
* Received at least 1L of fluid at ER entrance

Exclusion Criteria:

* Isolated head injury
* Isolated spine injury
* Chemotherapy within the last month
* Hematologic disease
* Chronic hemodialysis
* Uricase treatment within the last week
* Expected death within 48h

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Multiple trauma patients admitted in the trauma center and requiring ICU admission.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-09-30 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of serial plasmatic uric acid sampling after trauma | 7 days
  Number of measures collected/number of measures planned

SECONDARY OUTCOMES:
Impact of resuscitation on uric acid measures | 24 to 48 hours
  Impact of fluid administration (amount in mL) on the changes of subsequent uric acid blood level
Clinical predictors of the first blood uric acid (μmol/L) level measured | 12 hours
  Impact of patient's characteristics and physiological variables on the first measured blood uric acid.
  Characteristics will include: age (years), gender, Injury severity score, presence of acute renal impairment.
  Physiological variables will include: lower systolic blood pressure, base deficit, lactate level

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec, Canada